CLINICAL TRIAL: NCT04688411
Title: An mHealth Strategy to Improve Medication Adherence in Adolescents With Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sherif Badawy, MD, Assistant Professor, Department of Pediatrics, Division of Hematology, Oncology and Stem Cell Transplant, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 2020-3367; 1K23HL150232 (NIH)
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease; Sickle Beta Zero Thalassemia; Sickle B+ Thalassemia; Sickle Cell Hemoglobin C
Keywords: sickle cell disease; hydrxoyurea; mHealth intervention
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MED-Go app Intervention (Other): Participants will use MED-Go app intervention for a total of 12 weeks
  Interventions: Behavioral: MED-Go App
- Control Arm (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: MED-Go App — A novel multifunctional mobile app (MED-Go) to improve adherence to hydroxyurea in patients with sickle cell disease
  Arms: MED-Go app Intervention

SUMMARY:
The primary objective of this study is to evaluate a potential behavioral intervention (MED-Go app). To meet this objective, the researchers will conduct a pilot randomized controlled trial to test the feasibility and acceptability of MED-Go app in adolescents and young adults (AYA) with sickle cell disease (SCD). The long-term goal of this research is to promote medication adherence behavior and improve health outcomes in AYA with SCD.

DETAILED DESCRIPTION:
Sickle cell disease is the most common genetic disorder in the US, affecting about 100,000 Americans, and about 1 in 400 African American live births, incurring annual health care costs of $335 million. SCD can lead to serious complications including unpredictable, debilitating pain episodes, cardiopulmonary disease, stroke, and long-term end organ damage.These complications lead to significant declines in health-related quality of life (HRQOL) and other patient-reported outcomes (PROs), culminating in early mortality, particularly among AYA. Hydroxyurea (HU), at present, is the main FDA approved medication for SCD that reduces morbidity and mortality, improves HRQoL and lowers healthcare utilization.However, adherence to HU remains suboptimal with only 35-50% of patients achieving high adherence (≥90%), particularly among AYA with SCD. Low HU adherence has been associated with worse health outcomes, poor HRQOL and increased healthcare utilization. Low HU adherence is multifactorial, especially in AYA with other competing priorities and vulnerability in developmental and psychological factors contributing to adherence behavior. AYA have adopted text messaging and smartphone apps at a fast pace, including those who have SCD.Existing evidence indicates that mobile health (mHealth) behavioral interventions are feasible and acceptable with modest efficacy at improving medication adherence and self-management in AYA, including SCD. The specific aim for this study is to test the feasibility and acceptability of the MED-Go app as an mHealth behavioral intervention to improve HU adherence among AYA with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-21 years old
* Any sickle cell disease genotype
* On steady state of hydroxyurea for 2 months
* Own of have access to a smartphone during the study period

Exclusion Criteria:

* Recent hospitalizations within the past 7 days

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving feasibility criteria of using the MED-Go app | 12 weeks
  Feasibility is defined as 70% of participants logging their daily HU 70% of the time over 12 weeks or 59 out of 84 study days. This will be reported as a dichotomous outcome, either yes or no.

SECONDARY OUTCOMES:
Scores of System Usability Scale (SUS) | 12 weeks
  App usability questionnaires, numerical values, range 10-50 (higher scores indicating better usability of the app)
Hydroxyurea adherence rates | 12 weeks
  Adherence rate is defined as number of given HU doses as recorded by the app divided by total number of doses during study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M. Badawy, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
All patient data will be deidentified